CLINICAL TRIAL: NCT03510481
Title: Randomized, Placebo-Controlled, Double-Blind Study to Assess Safety, Immunogenicity, and Protective Efficacy of Two Regimens of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) During Natural Transmission Season in Healthy African Adults in Mali
Brief Title: Safety, Immunogenicity, and Protective Efficacy of Two Regimens of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) During Natural Transmission Season in Healthy African Adults in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanaria Inc. (Industry); Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999918084; 18-I-N084
Record Dates: First submitted 2018-04-26; First posted 2018-04-27 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-05

CONDITIONS: Malaria
Keywords: PfSPZ Vaccine; Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution; Artemether; Lumefantrine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Experimental arm 1: Dosing interval 0, 8, 16, and 54 weeks (Experimental): Participants received 3 doses of PfSPZ Vaccine (9 x 10^5) via direct venous inoculation (DVI) at 0, 8, 16 weeks and a 4th dose at 38 weeks post 3rd vaccination. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
  Interventions: Biological: PfSPZ Vaccine; Drug: artemether 20mg/lumefantrine 120mg (AL)
- Experimental arm 2: Dosing interval 0, 1, 4, and 42 weeks (Experimental): Participants received 3 doses of PfSPZ Vaccine (9 x 10^5) via direct venous inoculation (DVI) at 0, 1, 4 weeks and a 4th dose at 38 weeks post 3rd vaccination. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
  Interventions: Biological: PfSPZ Vaccine; Drug: artemether 20mg/lumefantrine 120mg (AL)
- Placebo comparator 3a: Dosing interval 0, 8, 16, and 54 weeks (Placebo Comparator): Control for Arm 1. Participants received 3 doses of placebo saline injection via direct venous inoculation (DVI) at 0, 8, 16 weeks and a 4th dose at 38 weeks post 3rd injection. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
  Interventions: Drug: Normal Saline; Drug: artemether 20mg/lumefantrine 120mg (AL)
- Placebo comparator 3b: Dosing interval 0, 1, 4, and 42 weeks (Placebo Comparator): Control for Arm 2. Participants received 3 doses of placebo saline injection via direct venous inoculation (DVI) at 0, 1, 4 weeks and a 4th dose at 38 weeks post 3rd injection. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
  Interventions: Drug: Normal Saline; Drug: artemether 20mg/lumefantrine 120mg (AL)

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ Vaccine is Radiation attenuated, aseptic, purified, vialed, cryopreserved, NF54 P. falciparum sporozoites produced by Sanaria, Inc.
  Arms: Experimental arm 1: Dosing interval 0, 8, 16, and 54 weeks; Experimental arm 2: Dosing interval 0, 1, 4, and 42 weeks
Drug: Normal Saline — Clear liquid indistinguishable from the study product will be used as a placebo rather than a comparator vaccine.
  Arms: Placebo comparator 3a: Dosing interval 0, 8, 16, and 54 weeks; Placebo comparator 3b: Dosing interval 0, 1, 4, and 42 weeks
Drug: artemether 20mg/lumefantrine 120mg (AL) — Licensed antimalarial in the US and Mali for use for uncomplicated malaria.
  Other Names: Coartem

SUMMARY:
Background:

The disease malaria affects many people in Mali and other parts of Africa and the world. It is caused by germs spread by mosquito bites. Malaria may be mild. But it can also be serious or lead to death if it is not treated promptly. Researchers want to find a safe vaccine that prevents malaria.

Objective:

To study how safe and tolerable the malaria vaccine called PfSPZ Vaccine is for healthy adults.

Eligibility:

Healthy adults:

* ages 18-35 in Ouelessebougou, Mali
* not infected with HIV, hepatitis B, or hepatitis C
* for females, not pregnant or breastfeeding and must use reliable birth control during the study

Design:

Participants will be screened with questions about malaria and will undergo blood, urine, and heart tests.

Participants will be randomly assigned to 1 of 4 groups. They will get injections of either the PfSPZ Vaccine or a salt-water placebo. They will not know which one they get.

Vaccinations will occur leading into the malaria transmission each year with 3 injections leading into Year 1 (malaria transmission season in 2018) and 1 injection prior to Year 2 (malaria transmission season 2019).

One vaccine group and one placebo group will get an injection 3 times over 4 weeks with an additional vaccination ~10 months later.

The other two groups (vaccine group and placebo) will get an injection 3 times over 16 weeks with an additional vaccination ~10 months later.

All participants will be treated with an antimalarial medication prior to the third injection and prior to fourth injection.

They will be followed for approximately 6 months after third and fourth injection.

At vaccine visits, female participants will have a pregnancy test before injection. All participants will have an arm cleaned and the vaccine injected in a vein. They will be watched for 30 minutes.

At non-vaccine visits, participants will have a physical exam and be asked how they are feeling. They will usually have blood tests.

DETAILED DESCRIPTION:
It is known that humans can be protected against malaria by repeated immunization with radiation-attenuated sporozoites. Sanaria, Inc. has developed a process for manufacturing, in compliance with current Good Manufacturing Practices (cGMPs) aseptic, purified, radiation- attenuated cryopreserved sporozoites from a well-characterized isolate of Plasmodium falciparum (Pf). This product, which is called PfSPZ Vaccine, can be administered by needle and syringe.

A collaboration among the Malaria Research and Training Center (MRTC, Mali), the Laboratory of Malaria Immunology and Vaccinology (LMIV) National Institute of Allergy and Infectious Diseases (NIAID), and Sanaria, Inc. has shown that sterile protection against naturally occurring malaria infection can be achieved. In this study, five doses of 2.7 x 10^5 PfSPZ during the dry season resulted in protective efficacies of about 48% by time to first positive blood smears (BS) and about 29% by proportion of participants with at least one positive BS during a full malaria transmission season (20 weeks), higher than those reported for other malaria vaccine candidates.

A follow up study in 2015 (ClinicalTrials.gov Identifier: NCT02627456) that reduced the number of vaccinations (from 5 to 3) while increasing the dose of sporozoites at each vaccination (2.7 x10^5 to 1.8x10^6 PfSPZ Vaccine) was conducted. Preliminary results show that 42 of 55 (77.8%) participants from the placebo group and 32 of 54 participants (58.1%) from the vaccine group developed Pf infection. Per protocol, the vaccine efficacy (VE) was 51% (p=0.004, 95% CI 20-70) by time-to-infection analysis (intention to treat (ITT) 39%, p=0.033) and 24% (p=0.031, 95% CI 2-41) by proportional analysis (ITT 22%, p= 0.041), similar to the previous study.

Studies are ongoing to establish a vaccination regimen, optimum dose and schedule, that will lead to improved sterile protection in endemic regions. Preliminary results from more recent studies in malaria-naïve and malaria-experienced participants have shown that 9.0x10^5 PfSPZ Vaccine dose per vaccination (lower than 1.8 x10^6 used in studies above) in a three-dose regimen may be an optimal dose for immunization. In addition, there is emerging evidence that a condensed, more practical regimen may also lead to development of sterile immunity. This proposed study is therefore designed to assess safety, immunogenicity and protective efficacy of two separate three-dose vaccination regimens during natural transmission season.

Participants in the main phase were randomized into arms receiving either PfSPZ Vaccine or normal saline injections. Each group received three doses of the respective injection during Year 1. After completion of the follow up in the main phase, all participants that are still enrolled in the study will be offered continued participation to receive a booster dose of the vaccine (dose # 4) with 9.0x10^5 PfSPZ or normal saline (depending on the group they were originally randomized to) at approximately 10 months post #3 vaccination. The booster dose is timed prior to ensuing malaria transmission season. Participants will be followed, similarly to the follow up during the main phase, for safety and vaccine efficacy for approximately 6 months during this second transmission season.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 and less than or equal to 35 years
  2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  3. In good general health and without clinically significant medical history
  4. Willing to have blood samples stored for future research
  5. Available for the duration of the study
  6. Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to Study Day 1 to 28 days after last vaccination.

     * Reliable methods of birth control include:

       * one of the following: confirmed pharmacologic contraceptives (parenteral) delivery; intrauterine or implantable device. OR
       * two of the following: a documented oral or transdermal or vaginal ring contraceptives; PLUS condoms with spermicide or diaphragm with spermicide.
     * Note, Coartem (artemether specifically) may reduce the effectiveness of systemic hormonal contraceptives, therefore additional barrier methods such as condoms must also be used during the 3 days of Coartem dosing.
     * Women who are not able to get pregnant will also be required to report date of last menstrual period, history of surgical sterility (i.e. tubal ligation, hysterectomy) or premature ovarian insufficiency (POI), and will have urine or serum pregnancy test performed per protocol.

EXCLUSION CRITERIA:

1. Pregnancy, as determined by a positive urine or serum human chorionic gonadotropin (beta-hCG) test (if female). NOTE: Pregnancy is also a criterion for discontinuation of any further dosing or non-safety related interventions for that subject.
2. Currently breast-feeding (if female)
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
4. Hemoglobin (Hb), WBC, absolute neutrophils, and platelets outside the local laboratory- defined limits of normal (subjects may be included at the investigator s discretion for not clinically significant values)
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal (subjects may be included at the investigator s discretion for not clinically significant values)
6. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B (HBV)
7. Known or documented sickle cell disease by history (Note: known sickle cell trait is NOT exclusionary)
8. Clinically significant abnormal electrocardiogram (ECG) such as abnormal QTc.
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
10. History of receiving any investigational product within the past 30 days
11. Participation or planned participation in a clinical trial with an investigational product prior to completion of the follow-up visit 28 days following last vaccination OR planned participation in an investigational vaccine study until the last required protocol visit
12. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
13. History of a severe allergic reaction(Grade 3 or higher or per PI discretion) or anaphylaxis
14. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that has required the use of oral or parenteral corticosteroids at any time during the past two years)
15. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia
16. Known immunodeficiency syndrome
17. Known asplenia or functional asplenia
18. Use of:

    * Chronic (greater than or equal to 14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of vaccination
    * Use of antimalarials or systemic antibiotics with known antimalarial activity within 5 drug half-lives prior to the first vaccine (such as artemether, artemether-lumefantrine, sulfadoxine-pyrimethamine, trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones or azithromycin)
19. Receipt of a live vaccine within the past four weeks or a killed vaccine within the past two weeks prior to Vaccination #1 and every subsequent vaccination day
20. Receipt of immunoglobulins and/or blood products within the past six months
21. Previous receipt of an investigational malaria vaccine in the last five years
22. Known allergies or other contraindications against Coartem
23. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 478 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Sissoko MS, Healy SA, Katile A, Omaswa F, Zaidi I, Gabriel EE, Kamate B, Samake Y, Guindo MA, Dolo A, Niangaly A, Niare K, Zeguime A, Sissoko K, Diallo H, Thera I, Ding K, Fay MP, O'Connell EM, Nutman TB, Wong-Madden S, Murshedkar T, Ruben AJ, Li M, Abebe Y, Manoj A, Gunasekera A, Chakravarty S, Sim BKL, Billingsley PF, James ER, Walther M, Richie TL, Hoffman SL, Doumbo O, Duffy PE. Safety and efficacy of PfSPZ Vaccine against Plasmodium falciparum via direct venous inoculation in healthy malaria-exposed adults in Mali: a randomised, double-blind phase 1 trial. Lancet Infect Dis. 2017 May;17(5):498-509. doi: 10.1016/S1473-3099(17)30104-4. Epub 2017 Feb 16. PMID 28216244
- [Background] Jongo SA, Church LWP, Mtoro AT, Schindler T, Chakravarty S, Ruben AJ, Swanson PA, Kassim KR, Mpina M, Tumbo AM, Milando FA, Qassim M, Juma OA, Bakari BM, Simon B, James ER, Abebe Y, Kc N, Saverino E, Fink M, Cosi G, Gondwe L, Studer F, Styers D, Seder RA, Schindler T, Billingsley PF, Daubenberger C, Sim BKL, Tanner M, Richie TL, Abdulla S, Hoffman SL. Increase of Dose Associated With Decrease in Protection Against Controlled Human Malaria Infection by PfSPZ Vaccine in Tanzanian Adults. Clin Infect Dis. 2020 Dec 31;71(11):2849-2857. doi: 10.1093/cid/ciz1152. PMID 31782768
- [Derived] Diawara H, Healy SA, Mwakingwe-Omari A, Issiaka D, Diallo A, Traore S, Soumbounou IH, Gaoussou S, Zaidi I, Mahamar A, Attaher O, Fried M, Wylie BJ, Mohan R, Doan V, Doritchamou JYA, Dolo A, Morrison RD, Wang J, Hu Z, Rausch KM, Zeguime A, Murshedkar T, Kc N, Sim BKL, Billingsley PF, Richie TL, Hoffman SL, Dicko A, Duffy PE; PfSPZ Vaccine Study Team. Safety and efficacy of PfSPZ Vaccine against malaria in healthy adults and women anticipating pregnancy in Mali: two randomised, double-blind, placebo-controlled, phase 1 and 2 trials. Lancet Infect Dis. 2024 Dec;24(12):1366-1382. doi: 10.1016/S1473-3099(24)00360-8. Epub 2024 Aug 14. PMID 39153490

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 478 subjects signed consent. 251 subjects were screen failures. 17 subjects were enrolled but not vaccinated. 210 subjects started the study.
Groups:
- Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks: Participants received 3 doses of PfSPZ Vaccine (9 x10^5) via direct venous inoculation (DVI) at 0, 8, 16 weeks and a 4th dose at 38 weeks post 3rd vaccination. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
- Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks: Participants received 3 doses of PfSPZ Vaccine (9 x10^5) via direct venous inoculation (DVI) at 0, 1, 4 weeks and a 4th dose at 38 weeks post 3rd vaccination. Oral antimalarial treatment with artemether 20mg/lumefantrine 120mg (AL) given orally with food with 4 tablets taken as a single initial dose, then 4 tabs again after 8hrs, then 4 tabs twice daily for the following two days for a total of 24 tabs, 2 weeks prior to 3rd and 4th injection.
Period: Year 1
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks
Started | 69 | 70 | 36 | 35
Completed | 56 | 61 | 34 | 31
Not Completed | 13 | 9 | 2 | 4
Period: Year 2 - Booster Dose
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks
Started | 46 (10 participants who completed Period 1 did not re-consent for Period 2.) | 52 (9 participants who completed Period 1 did not re-consent for Period 2.) | 25 (9 participants who completed Period 1 did not re-consent for Period 2.) | 19 (12 participants who completed Period 1 did not re-consent for Period 2.)
Completed | 42 | 49 | 23 | 18
Not Completed | 4 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks | Total
Number analyzed (Participants) | 69 | 70 | 36 | 35 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 70 | 36 | 35 | 210
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 31 | 10 | 13 | 74
  Male | 49 | 39 | 26 | 22 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Bambara | 48 | 43 | 25 | 18 | 134
  Bozo | 0 | 0 | 0 | 1 | 1
  Malinke | 5 | 8 | 2 | 5 | 20
  Peuhl | 3 | 7 | 4 | 2 | 16
  Sarakole | 6 | 2 | 2 | 1 | 11
  Songrai | 3 | 2 | 0 | 0 | 5
  Other | 4 | 8 | 3 | 8 | 23
Region of Enrollment [Number; unit: participants]
  Mali | 69 | 70 | 36 | 35 | 210

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events in Year One
Description: Incidence of local and systemic adverse events (AEs) graded by severity occurring within 7 days after each vaccine administration in year one
Time Frame: Within 7 days after each vaccination in year one
Population: The analyses included only subjects who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks
Number analyzed (Participants) | 69 | 70 | 36 | 35
Participants | 39 | 27 | 19 | 11

2. Primary Outcome: Number of Participants With Local and Systemic Adverse Events in Year Two
Description: Incidence of local and systemic adverse events (AEs) graded by severity occurring within 7 days after vaccine administration during year two (booster dose)
Time Frame: Within 7 days after each vaccination in year two
Population: The analyses included only subjects who received fourth dose of vaccine in year two
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks
Number analyzed (Participants) | 46 | 52 | 25 | 19
Participants | 5 | 12 | 3 | 2

ADVERSE EVENTS:
Time Frame: For the primary endpoint, other (non-serious) adverse events were monitored 7 days from time of each vaccination during year one and year two. Deaths and serious AEs were monitored up to 21 months (duration of the study).
Arm/Group | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70 | 1/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/69 | 0/70 | 1/36 | 0/35
Other Adverse Events (participants affected / at risk) | 41/69 | 34/70 | 20/36 | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks (N=69) | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks (N=70) | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks (N=36) | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks (N=35)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm 1: Dosing Interval 0, 8, 16, and 54 Weeks (N=69) | Experimental Arm 2: Dosing Interval 0, 1, 4, and 42 Weeks (N=70) | Placebo Comparator 3a: Dosing Interval 0, 8, 16, and 54 Weeks (N=36) | Placebo Comparator 3b: Dosing Interval 0, 1, 4, and 42 Weeks (N=35)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 3 (3) | 3 (3) | 4 (5) | 2 (2)
CHILLS (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
GRANULOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 13 (14) | 14 (16) | 6 (7) | 3 (3)
HEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 7 (7) | 7 (8) | 7 (7) | 4 (4)
MALAISE (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 11 (13) | 8 (8) | 6 (7) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (3) | 3 (4) | 3 (6) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
NIAID cannot contact the FDA regarding the trial independent of the IND Sponsor (Sanaria, Inc.).

Dr. Patrick Duffy is employed by the clinical sponsor, NIAID (clinical sponsor). Dr. Diawara is not employed by either sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03510481/Prot_SAP_000.pdf